CLINICAL TRIAL: NCT04661332
Title: Registro Delle Colangiopancreatografie Retrograde Endoscopiche Eseguite in Humanitas
Brief Title: Registry of Endoscopic Retrograde Cholangiopancreatographies Performed in Humans
Acronym: ERCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2143
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: ERCP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic retrograde cholangio-pancreatography: Endoscopic retrograde cholangio-pancreatography procedure

SUMMARY:
Treatment of the pathology of the extrahepatic biliary tract is the most frequent indication for performing endoscopic retrograde cholangiography (ERCP). The method, which combines endoscopic and radiological vision, also allows for therapeutic (and diagnostic) procedures on some pathologies of the pancreas and the papilla of Vater.

During the maneuvers it is also possible to obtain cyto-histological material for the diagnosis of any lesions identified, through the execution of brushing.

The endoscope used for ERCP allows for microsurgical procedures to be performed on the papilla of Vater, on the biliary tract and on the pancreas, procedures that in the past required a real surgical intervention.

ERCP is a generally well tolerated procedure, but as with all medical procedures it can have limitations and be followed by some complications. In 5% of cases, the procedure may not be completed due to anatomical variants that do not allow the endoscope to reach the duodenum or to cannulate and visualize the bile and / or pancreatic ducts. The most frequent complication is acute pancreatitis, which can arise as a consequence of surgery on the common outlet of the biliary and pancreatic tracts; it occurs in 3-5% of cases and to date, it cannot be predicted or prevented in all cases. In some groups of patients (young, with non-dilated biliary tract, or with a history of previous pancreatitis) the risk of pancreatitis can reach 10-12% . In rare cases (less than 1%), pancreatitis can have a severe course and may require surgery. Other less frequent complications (with an overall incidence of less than 2%) are: infection of the biliary tract or cystic collections, bleeding resulting from papillo-sphincterotomy, and perforation of the duodenum or ducts. Infection and bleeding are generally treated medically or endoscopically; the perforation may require surgery in some cases.

This registry aims to collect in a prospective and / or retrospective way the data of the ERCP procedures performed in our center by evaluating the sex, age of the patient, the reason why the patient was subjected to the examination, diagnosis, clinical risk factors and technical risk (i.e. associated with the procedure itself), if there have been complications, the type of instrumentation in use in our operating unit and / or the operators performing the examinations.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be recruited at the ICH Gastroenterology and Digestive Endoscopy Unit. The patients in question will be subjects of both sexes, over the age of 18 and who need to undergo ERCP.

Exclusion Criteria:

* Patients under 18 or unable to express informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited at the ICH Gastroenterology and Digestive Endoscopy Unit. The patients in question will be subjects of both sexes, over the age of 18 and who need to undergo ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To collect the information of all the ERCPs performed in the hospital | 10 years
  This study aims to collect the information of all the ERCPs performed in the hospital in order to know the current clinical practice in order to identify any margins for improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: No